CLINICAL TRIAL: NCT06494852
Title: Association of Renal-tubular Acidosis in Children With Cow Milk Protein Allergy
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Esraa Mohamed Hedia, MBBCh, Sohag University
Other Study IDs: Soh-Med-24-5-02MS
Record Dates: First submitted 2024-07-02; First posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Cow's Milk Protein Allergy; Rta
Keywords: CMPA / RTA
MeSH Terms: conditions — Milk Hypersensitivity; Acidosis, Renal Tubular | interventions — Physical Examination

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: investigations — laboratory assesment Kidney function test, Urine analysis, Arterial blood gases ,Electrolytes (Na,K,Cl,Ca,phosphorus) and Calcium/creatinine ratio , Total serum IgE Radiological assessment Abdominal ultrasonography

SUMMARY:
Our study aims to detect renal manifestations of children proved to be with cow milk protein allergy special focusing on tubular dysfunction.

DETAILED DESCRIPTION:
This is a cross-sectional study that will be conducted over 6 months at the pediatric department, Sohag University Hospital, Sohag, Egypt.

Children proved to be with cow milk protein allergy by oral challenge test after stabilization and prevention of cow protein with Age group from 3 months up to 3 years attending outpatient clinic at Sohag University Hospital will be included in the study.

The study participants will be subjected to full history taking and thorough clinical examination at the pediatric outpatient clinic and their medical files will be reviewed.

ELIGIBILITY:
Inclusion Criteria:

* Children proved to be with cow milk protein allergy by oral challenge test after stabilization and prevention of cow protein with Age group from 3 months up to 3 years attending outpatient clinic at Sohag University Hospital will be included in the study

Exclusion Criteria:

-

Ages: 3 Months to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children proved to be with cow milk protein allergy by oral challenge test after stabilization and prevention of cow protein with Age group from 3 months up to 3 years
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2023-06-03 (Actual); Primary Completion 2023-12-03 (Actual); Study Completion 2024-01-03 (Actual)

PRIMARY OUTCOMES:
investigate association of Renal tubular acidosis in cow milk protein allergy patients | 6 months
  Our study aims to detect renal manifestations of children proved to be with cow milk protein allergy special focusing on tubular dysfunction

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
not decided yet if i will share my IPD or not